CLINICAL TRIAL: NCT02699125
Title: A Placebo Controlled Double Blinded Crossover Study of the Antihypertensive Efficacy of Guanfacine vs Hydrochlorothiazide in Obstructive Sleep Apnea (OSA) Associated Hypertension
Brief Title: Treatment of OSA Associated Hypertension With Alpha 2 Agonist or Diuretic
Acronym: guanhctz
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Michael G. Ziegler, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: guanhctz
Record Dates: First submitted 2016-02-26; First posted 2016-03-04 (Estimated); Results first posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Guanfacine; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo, Guanfacine, Hydrochlorothyazide (Experimental): Sequence: Placebo, Then Guanfacine1 mg for 2 weeks followed by guanfacine 2 mg for 4 weeks, Then Hydrochlorothiazide 12.5 mg for 2 weeks followed by hydrochlorothiazide 25 mg for 4 weeks.
  Interventions: Drug: Guanfacine; Drug: Hydrochlorothiazide
- Placebo, Hydrochlorothyazide, Guanfacine (Experimental): Sequence: Placebo, Then Hydrochlorothiazide 12.5 mg for 2 weeks followed by hydrochlorothiazide 25 mg for 4 weeks, Then Guanfacine1 mg for 2 weeks followed by guanfacine 2 mg for 4 weeks.
  Interventions: Drug: Guanfacine; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Guanfacine — Guanfacine 1mg for 2 weeks followed by guanfacine 2mg for 4 weeks.
  Other Names: Tenex
Drug: Hydrochlorothiazide — Hydrochlorothiazide 12.5 mg for 2 weeks followed by hydrochlorothiazide 25 mg for 4 weeks
  Other Names: Hydrodiuril

SUMMARY:
Patients who have obstructive sleep apnea (OSA) frequently stop breathing while they sleep. They often develop high blood pressure. We are not sure what drug is best to treat the high blood pressure. This study will give the patients guanfacine or hydrochlorothiazide (HCTZ) for 6 weeks after 2 weeks of placebo. The blood pressure response will be evaluated by 24 hour monitoring.

DETAILED DESCRIPTION:
This is a blinded crossover study measuring the antihypertensive efficacy of guanfacine vs HCTZ in up to 34 subjects. Subjects with an apnea-hypopnea index (AHI) > 10 and hypertension can enter the study. Hypertension is defined as a systolic blood pressure (SBP) > 140 or a diastolic blood pressure (DBP) > 90 on the average of three seated blood pressure measurements or a history of medical therapy for hypertension. Subjects who have tried and abandoned continuous positive airway pressure (CPAP) therapy for sleep apnea are eligible for this study. All others will be advised that CPAP is preferred treatment for sleep apnea and are eligible only if they decline CPAP or use it for too short a time at night to be effective.

Then patients will have their antihypertensive drugs tapered off and receive single blind placebo for two weeks. After that, all subjects receive guanfacine or HCTZ for six weeks with a full evaluation at that time. Subjects are crossed over to HCTZ 12.5 mg for 2 weeks followed by HCTZ 25 mg for 4 more weeks Guanfacine 1mg will be taken daily at bedtime for 2 weeks and then as a dose of 2 mg for the remaining 4 weeks. Subjects will receive a telephone call at the time of increased dosage as a reminder. Blood, urine and 24-hour blood pressure measurements, hemodynamic measurements, questionnaires and drug accountability are measured in the same manner toward at the the end of placebo and each drug treatment. The entire study will take 14 weeks, although each study period may be lengthened by one week if necessary for the convenience of the subject's personal schedule.

Patients will provide blood pressure readings from their home monitor or in clinic and will not have the dose increased if they have systolic blood pressure below 105 mm Hg or side effects, such as excessive somnolence, drowsiness, or depression, suggesting that an increased dose might worsen side effects

At the end of each treatment period, subjects will undergo noninvasive hemodynamic testing. Ultrasound will be used to measure aortic diameter and blood velocity in the ascending aorta in order to better estimate cardiac output. Then, finger plethysmography will be used to acquire beat-to-beat finger blood pressure and pulse rate. Beat-to-beat derived hemodynamic variables will be calculated by a model flow algorithm (e.g. brachial artery flow, stroke volume, cardiac output, ejection time, blood pressure rate of change, peripheral resistance). Applanation tonometry will be used to obtain pulse wave velocity and central arterial pressure. ECG will be recorded with standard ECG leads to determine heart rate variability in both time and frequency domains. Spontaneous baroreflex will be determined from beat-to-beat changes in blood pressure and pulse pressure interval. Forearm reactive hyperemia will be used to quantify endothelial dysfunction during 4 minutes of post-ischemic change. Subjects will then complete an Epworth Sleepiness Scale questionnaire (ESS) and a Functional Outcomes of Sleep Questionnaire (FOSQ) to find whether they are drowsy in the daytime and if they feel that they are compromised by not having adequate rest. Any adverse event will be recorded. They are asked about any concurrent medication over the prior period, including prescription medication, over the counter medication, and caffeine intake. Medication compliance is evaluated by pill count. Those who fail to return their pill bottle are requested to bring it in. Finally, a 24-hour ambulatory blood pressure monitor (ABPM) will be attached to automatically collect blood pressure and heart rate values every 15 minutes during the wake period and every 30 minutes during the sleep period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ranging from 20 - 80 years
2. Body mass index (BMI) of 20-38 to include the typical obese OSA patients and avoid the practical difficulties in blood drawing from the massively obese
3. Hypertension with blood pressures > 140/90 but less than 180/105 mmHg.
4. Apnea-hypopnea index above 10

Exclusion Criteria:

1. Receiving medications other than anti-hypertensives known to influence the sympathetic nervous system, sleep medicines (including heavy alcohol use) or drugs with adverse interactions with study medication.
2. Women who have premenstrual syndrome, or those who are pregnant or capable of pregnancy and unwilling to use effective non-hormonal contraception
3. Shift workers or have symptoms of narcolepsy, restless legs syndrome or insomnia, in order to minimize confounding effects of other sleep disorders
4. Have apneas which are primarily central
5. Have sleep fragmentation caused by syndromes such as chronic pain or movement disorders
6. Have diseases such as asthma or chronic obstructive pulmonary disease that compromises respiration.
7. Have known coronary or cerebral vascular disease, history of arrhythmias, cardiomyopathy, history of psychosis, current alcohol or drug abuse.
8. Have any contraindications to any study materials, such as heart block.
9. Have secondary hypertension
10. Have creatinine levels above 2.5 mg %, more than 1+ proteinuria by dipstick, hematuria or electrolyte disorders.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael G. Ziegler, M.D., Principal Investigator — UCSD

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ziegler MG, Milic M, Sun P. Antihypertensive therapy for patients with obstructive sleep apnea. Curr Opin Nephrol Hypertens. 2011 Jan;20(1):50-5. doi: 10.1097/MNH.0b013e3283402eb5. PMID 21326007
- [Derived] Ziegler MG, Milic M, Dimsdale JE, Mills PJ. Sympathetic overactivity and nocturnal diuresis in obstructive sleep apnea alter the response to hypertension therapy. Clin Hypertens. 2024 Jun 1;30(1):14. doi: 10.1186/s40885-024-00272-x. PMID 38822391

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 405 participants were screened for eligibility.
Pre-assignment Details: 41 participant was enrolled in the study.
Groups:
- Placebo, Then Guanfacine, Then Hydrochlorothiazide: Participants first received Placebo for 2 weeks. They then received guanfacine 1 mg for 2 weeks followed by guanfacine 2 mg for 4 weeks. They then received hydrochlotothyazide 12.5 mg for 2 weeks followed by hydrochlorothyazied 25 mg for 4 weeks.
- Placebo, Then Hydrochlorothiazide Then Guanfacine.: Participants first received Placebo for 2 weeks. They then received hydrochlotothyazide 12.5 mg for 2 weeks followed by hydrochlorothyazied 25 mg for 4 weeks. They then received guanfacine 1 mg for 2 weeks followed by guanfacine 2 mg for 4 weeks.
Period: Placebo
Arm/Group | Placebo, Then Guanfacine, Then Hydrochlorothiazide | Placebo, Then Hydrochlorothiazide Then Guanfacine.
Started | 21 | 20
Completed | 18 | 16
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 4
Period: First Intervention (6 Weeks).
Arm/Group | Placebo, Then Guanfacine, Then Hydrochlorothiazide | Placebo, Then Hydrochlorothiazide Then Guanfacine.
Started | 18 | 16
Completed | 18 | 16
Not Completed | 0 | 0
Period: Second Intervention (6 Weeks).
Arm/Group | Placebo, Then Guanfacine, Then Hydrochlorothiazide | Placebo, Then Hydrochlorothiazide Then Guanfacine.
Started | 18 | 16
Completed | 11 | 14
Not Completed | 7 | 2
Not completed — Withdrawal by Subject | 7 | 2

BASELINE CHARACTERISTICS:
Population: Analyzed Baseline population for the primary outcome (21) and secondary outcome (18) is not consistent with the Overall Number of Baseline (Placebo) Participants (34) in the Participant Flow Module because (13) and (16) participants respectfully were excluded from the analysis due to either missing data and/or low quality ultrasound images.
Groups:
- Placebo: "Placebo" column have 6 rows of baseline Primary Outcome Values: "24-h", "Wake" and "Sleep" Systolic and Diastolic Blood Pressure. "Placebo" column also have 1 row of baseline Secondary Outcome Value: Brachial Artery Flow Mediated Dilation.
Arm/Group | Placebo
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 21
24-h, Wake and Sleep Period Systolic and Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Systolic Blood Pressure and Distolic Blood Pressure recorded during the Overall 24-h Period, every 15 minutes during the Wake Period and every 30 minutes during the Sleep Period.
  mmHg
    24-h systolic blood pressure | 143 (19)
    24-h diastolic blood pressure | 87 (11)
    Wake systolic blood pressure | 147 (20)
    Wake diastolic blood pressure | 91 (12)
    Sleep systolic blood pressure | 136 (20)
    Sleep diastolic blood pressure | 80 (11)
Brachial Artery Flow Mediated Dilation [Mean (Standard Deviation); unit: percent] — Brachial Artery Flow Mediated Dilation is the maximal right brachial artery dilation during the reactive hyperemia following the release of the 5-minute cuff occlusion of the right forearm. Population: The Overall Number of Participants Analyzed (18) differs from the Overall Number of Baseline Participants (21) because brachial artery flow mediated dilation data for 3 participants were excluded due to low quality of the ultrasound images.
  percent
    number analyzed (Participants) | 18
    (all) | 4.5 (3)

OUTCOME MEASURES:

1. Primary Outcome: 24-h, Wake and Sleep Period Systolic and Diastolic Blood Pressure
Description: The primary outcome measure is ambulatory systolic and diastolic blood pressure recorded once every 15 minutes during the day and once every 30 minutes during the sleep. The Outcome Measure Data Table present primary outcome as "24-h", "Wake" and "Sleep" Period Systolic and Diastolic Blood Pressure after each of the following three interventions: Placebo, Guanfacine and Hydrochlorothiazide.
Time Frame: At the end of 2 weeks of placebo therapy, at the end of 6 weeks of guanfacine therapy and at the end of 6 weeks of hydrochlorothiazide therapy.
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Placebo: Placebo for 2 weeks
- Guanfacine: Guanfacine 1 mg for 2 weeks followed by guanfacine 2 mg for 4 weeks.
- Hydrochlorothyazide: Hydrochlorothyazide 12.5 mg for 2 weeks followed by hydrochlorothyazide 25 mg for 4 weeks.
Arm/Group | Placebo | Guanfacine | Hydrochlorothyazide
Number analyzed (Participants) | 21 | 21 | 21
mmHg
  24-h systolic blood pressure | 143 (4.2) | 133 (2.9) | 136 (3.5)
  24-h diastolic blood pressure | 87 (2.5) | 81 (2) | 83 (2.3)
  Wake systolic blood pressure | 147 (4.4) | 137 (3.1) | 139 (3.9)
  Wake diastolic blood pressure | 91 (2.7) | 84 (1.9) | 86 (2.5)
  Sleep systolic blood pressure | 136 (4.3) | 124 (2.6) | 130 (3.4)
  Sleep diastolic blood pressure | 80 (2.4) | 73 (2.3) | 76 (2.3)

2. Secondary Outcome: Brachial Artery Flow Mediated Dilation
Description: Brachial Artery Flow Mediated Dilation is upper arm brachial artery dilation during the 3 minutes forearm reactive hyperemia following the release of the 5-minute forearm cuff occlusion.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of the preoclussion diameter
Groups:
- Hydrochlorothiazide: Hydrochlorothyazide 12.5 mg for 2 weeks followed by hydrochlorothyazide 25 mg for 4 weeks.
Arm/Group | Placebo | Guanfacine | Hydrochlorothiazide
Number analyzed (Participants) | 18 | 18 | 18
percentage of the preoclussion diameter | 4.5 (0.8) | 8.4 (1.1) | 4.9 (0.7)

ADVERSE EVENTS:
Time Frame: 14 Weeks
Arm/Group | Placebo | Guanfacine | Hydrochlorothiazide
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No